CLINICAL TRIAL: NCT07228403
Title: A 104-week, Multicenter, Open-label, Single-arm, Phase 3 Extension Trial Investigating the Long-term Safety and Efficacy of Glepaglutide in Adult Patients With Short Bowel Syndrome (SBS) Rolling Over From the EASE SBS 2 or 3 Trials
Brief Title: Efficacy and Safety Evaluation of Glepaglutide in Treatment of Short Bowel Syndrome
Acronym: EASE SBS 6
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZP1848-25009; 2025-520775-81-00 (EU CTIS Number); U1111-1317-8307 (Other: UT Number)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Short Bowel Syndrome (SBS)
Keywords: Malabsorption Syndromes; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Postoperative Complications; Pathologic Processes; Pathological Conditions, Signs and Symptoms; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome; Malabsorption Syndromes; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Postoperative Complications; Pathologic Processes; Pathological Conditions, Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label Glepaglutide (Experimental)
  Interventions: Drug: Glepaglutide 10 mg

INTERVENTIONS:
Drug: Glepaglutide 10 mg — Administered twice weekly by subcutaneous injection for a maximum of 24 months
  Other Names: ZP1848

SUMMARY:
The purpose of this study is to understand the safety and efficacy of twice weekly glepaglutide 10 mg in adult patients with short bowel syndrome (SBS), who were previously enrolled in the EASE SBS 2 or EASE SBS 3 trials. Participants currently on these trials will be able to continue their glepaglutide treatment by enrolling in this EASE SBS 6 extension trial. The trial includes a 24-month treatment period, followed by a 4-week safety follow-up period. Participants will attend trial visits, where they may undergo heart tests (electrocardiogram (ECG)), vital sign checks, colonoscopies, blood and urine tests, and physical exams.

DETAILED DESCRIPTION:
This trial is a 104-week, multicenter, open-label, single-arm, phase 3 extension trial investigating the long-term safety and efficacy of glepaglutide in adult patients with short bowel syndrome (SBS) rolling over from the EASE SBS 2 or 3 trials.

ELIGIBILITY:
Inclusion Criteria:

* Has provided signed informed consent and agrees to comply with protocol requirements.
* Is being

  1. Actively treated and has completed at least 6 months of glepaglutide treatment in the EASE SBS 2 trial, or
  2. Actively treated in the EASE SBS 3 trial.

Exclusion Criteria:

* Has a condition, disease, or circumstance that, in the opinion of the investigator, would put the patient at any undue risk, prevent completion of the trial, or confound the planned assessments of the trial.
* Use of GLP-1, GLP-2 (e.g., teduglutide), HGH, DPP-4 inhibitors, somatostatin, or analogs thereof. Note: Prior use of glepaglutide is allowed.
* Had major protocol deviation(s) (as determined by the sponsor) in the EASE SBS 2 or EASE SBS 3 trial that would affect the conduct of the present trial.
* Has permanently discontinued the trial treatment because of an AE, assessed as related to the trial drug in the EASE SBS 2 or EASE SBS 3 trial. (Note: AEs are treatment-emergent unless otherwise specified.)
* If female, is of childbearing potential, pregnant, breastfeeding, intends to become pregnant, or is not using contraceptive methods. Refer to Section 10.2.2 for the definition of contraception.
* Has a known or suspected hypersensitivity to glepaglutide or related products.
* Has committed to an institution by virtue of an order issued by the judicial or administrative authorities.
* Is an employee of the sponsor or investigator or otherwise dependent on them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2028-09-18 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From baseline to the safety follow-up visit (A maximum of 25 months)

SECONDARY OUTCOMES:
Change in prescribed weekly parenteral support (PS) volume | From baseline to Month 24 (End of Trial)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (4):
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Lied Transplant Center at Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic-9500 Euclid Ave, Cleveland, Ohio
  - Vanderbilt University Medical Center-Tennesse-1211 21st Ave S, Nashville, Tennessee
- UZ Leuven - PPDS, Leuven, Belgium
- LHSC - University Hospital, London, Ontario, Canada
- AP-HP - Hôpital Beaujon, Clichy, Hauts-de-Seine, France
- Germany (5):
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-Vorpommern
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin
  - Asklepios Klinik St. Georg, Hamburg
- Poland (3):
  - Szpital Skawina sp. z o.o. im. Stanley Dudricka, Skawina, Lesser Poland Voivodeship
  - Samodzielny Publiczny Szpitala Kliniczny im. Prof. Witolda Orlowskiego CMKP, Warsaw, Masovian Voivodeship
  - Wojewódzki Szpital Specjalistycznyo im. M. Pirogowa w Lodzi, Lodz
- St Mark's Hospital (Central Middlesex Hospital), Ealing, United Kingdom

IPD SHARING:
Plan to Share IPD: No